CLINICAL TRIAL: NCT02554656
Title: VFEND SPECIAL INVESTIGATION- INVESTIGATION FOR TREATMENT OF INVASIVE FUNGAL INFECTIONS IN PEDIATRIC PATIENTS -
Brief Title: Vfend Special Investigation For Pediatric - Observational
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501100
Record Dates: First submitted 2015-07-15; First posted 2015-09-18 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Safety and Effectiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Examine the safety and effectiveness of Vfend [voriconazole] for pediatric under general clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is under 15 years old and deep mycosis infection.

Exclusion Criteria:

* Patients who have been previously enrolled in this study. -

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subjects who have been treated with voriconazole for severe mycosis
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- XXXXXXX, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501100&StudyName=Vfend%20Special%20Investigation%20For%20Pediatric

RESULTS

PARTICIPANT FLOW:
Groups:
- VFEND (Voriconazole): Participants who received VFEND as indicated in the approved local product document were observed for a period of 16 weeks at maximum. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | VFEND (Voriconazole)
Started | 89
Completed | 86
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: A total of 89 participants were enrolled in this study. Of the 89 participants, 3 participants were excluded from the safety analysis set due to the following reason: Protocol violation (registration violation: 1, out of the study period: 2)
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 86
Age, Customized [Number; unit: Participants]
  <1 month after birth | 0
  ≥1 month and <1 year | 1
  ≥1 to <7 years | 40
  ≥7 to <15 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diagnostic Name (Name of Infection) [Number; unit: Participants] — Diagnosis name (name of infection) include definitive diagnosis and suspected cases.
  Participants
    Invasive aspergillosis | 34
    Pulmonary aspergilloma | 6
    Chronic necrotic pulmonary aspergillosis | 1
    Candidemia | 7
    Esophageal candidiasis | 2
    Candida peritonitis | 0
    Bronchopulmonary candidiasis | 2
    Cryptococcal meningitis | 0
    Pulmonary cryptococcosis | 0
    Fusariosis | 0
    Scedosporiosis | 0
    Other invasive fungal infections | 20
    Invasive fungal infections (multiple infections) | 2
    Other than invasive fungal infections | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to VFEND was assessed by the physician.
Time Frame: 16 weeks at maximum
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received VFEND at least once.
Measure: Number; unit: Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 86
Participants
  ADRs | 23
  Serious ADRs | 3

2. Secondary Outcome: Number of Participants With Adverse Drug Reactions Not Expected From the LPD (Unknown Adverse Drug Reaction)
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to VFEND was assessed by the physician.
Time Frame: 16 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 86
Participants | 2

3. Secondary Outcome: Incidence of Aadverse Reactions by Diagnosis (Infection)
Description: An ADR was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. Relatedness to VFEND was assessed by the physician. Participants with ADRs were counted by diagnosis (infection) to assess whether it was a risk factor for the occurrence of ADRs.
Time Frame: 16 weeks at maximum
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 86
Percentage of Participants
  Invasive aspergillosis: number analyzed (Participants) | 34
  Invasive aspergillosis | 35.29 [19.746 to 53.511]
  Pulmonary aspergilloma: number analyzed (Participants) | 6
  Pulmonary aspergilloma | 33.33 [4.327 to 77.722]
  Chronic necrotic pulmonary aspergillosis: number analyzed (Participants) | 1
  Chronic necrotic pulmonary aspergillosis | 100.00 [2.500 to 100.000]
  Candidemia: number analyzed (Participants) | 7
  Candidemia | 0.00 [0.000 to 40.962]
  Esophageal candidiasis: number analyzed (Participants) | 2
  Esophageal candidiasis | 0.00 [0.000 to 84.189]
  Candida peritonitis: number analyzed (Participants) | 0
  Bronchopulmonary candidiasis: number analyzed (Participants) | 2
  Bronchopulmonary candidiasis | 50.00 [1.258 to 98.742]
  Cryptococcal meningitis: number analyzed (Participants) | 0
  Pulmonary cryptococcosis: number analyzed (Participants) | 0
  Fusariosis: number analyzed (Participants) | 0
  Scedosporiosis: number analyzed (Participants) | 0
  Other invasive fungal infections: number analyzed (Participants) | 20
  Other invasive fungal infections | 20.00 [5.733 to 43.661]
  Invasive fungal infections (multiple infections): number analyzed (Participants) | 2
  Invasive fungal infections (multiple infections) | 50.00 [1.258 to 98.742]
  Other than invasive fungal infections: number analyzed (Participants) | 12
  Other than invasive fungal infections | 16.67 [2.086 to 48.414]

4. Secondary Outcome: Overall Clinical Response
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Overall clinical effectiveness of VFEND was assessed as "effective", "not effective", or "indeterminate" by the physician based on the clinical course at the end of the observation period or at the time of treatment discontinuation.
Time Frame: 16 weeks at maximum
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation at the end of the observation period or at the time of treatment discontinuation. The efficacy analysis sets were 74 participants. Participants assessed as "indeterminate (n=7)" at the final observation were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Parcentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 67
Parcentage of Participants | 80.6 [69.11 to 89.24]

5. Secondary Outcome: Clinical Response Rate by Diagnostic Name (Name of Infection)
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Overall clinical effectiveness of VFEND was assessed as "effective", "not effective", or "indeterminate" by the physician based on the clinical course at the end of the observation period or at the time of treatment discontinuation. Overall effectiveness of VFEND was determined by the physician based on the clinical course. Participants achieved clinical effectiveness by Diagnosis (Infection) were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 16 weeks at maximum
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 67
Percentage of Participants
  Invasive aspergillosis: number analyzed (Participants) | 33
  Invasive aspergillosis | 97.0 [84.24 to 99.92]
  Pulmonary aspergilloma: number analyzed (Participants) | 4
  Pulmonary aspergilloma | 75.0 [19.41 to 99.37]
  Chronic necrotic pulmonary aspergillosis: number analyzed (Participants) | 1
  Chronic necrotic pulmonary aspergillosis | 0.0 [0.00 to 97.50]
  Candidemia: number analyzed (Participants) | 5
  Candidemia | 100.0 [47.82 to 100.00]
  Esophageal candidiasis: number analyzed (Participants) | 2
  Esophageal candidiasis | 100.0 [15.81 to 100.00]
  Candida peritonitis: number analyzed (Participants) | 0
  Bronchopulmonary candidiasis: number analyzed (Participants) | 1
  Bronchopulmonary candidiasis | 100.0 [2.50 to 100.00]
  Cryptococcal meningitis: number analyzed (Participants) | 0
  Pulmonary cryptococcosis: number analyzed (Participants) | 0
  Fusariosis: number analyzed (Participants) | 0
  Scedosporiosis: number analyzed (Participants) | 0
  Other invasive fungal infections: number analyzed (Participants) | 19
  Other invasive fungal infections | 47.4 [24.45 to 71.14]
  Invasive fungal infections (multiple infections): number analyzed (Participants) | 2
  Invasive fungal infections (multiple infections) | 100.0 [15.81 to 100.00]

ADVERSE EVENTS:
Time Frame: 16 weeks at maximum
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | VFEND (Voriconazole)
All-Cause Mortality (participants affected / at risk) | 6/86
Serious Adverse Events (participants affected / at risk) | 11/86
Other Adverse Events (participants affected / at risk) | 41/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VFEND (Voriconazole) (N=86)
Cytomegalovirus viraemia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 1
Cytokine storm (Immune system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Pyrexia (General disorders) | 1
Lymphocyte count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VFEND (Voriconazole) (N=86)
Photophobia (Eye disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 3
Aspartate aminotransferase increased (Investigations) | 13
Alanine aminotransferase increased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 13
Platelet count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02554656/SAP_000.pdf
  • Study Protocol (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02554656/Prot_001.pdf